CLINICAL TRIAL: NCT07051486
Title: A Single-Arm, Multicenter Phase II Clinical Trial of SHR-A1811 for Injection in Patients With HER2-Expressing Recurrent or Metastatic Cervical Cancer Progressing After Standard Treatment
Brief Title: A Phase II Trial of SHR-A1811 in HER2-Expressing Recurrent/Metastatic Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-218
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Recurrent or Metastatic Cervical Cancer
MeSH Terms: conditions — Recurrence; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 Group (Experimental)
  Interventions: Drug: SHR-A1811 Injection

INTERVENTIONS:
Drug: SHR-A1811 Injection — SHR-A1811 for injection.

SUMMARY:
This study is a single-arm, multicenter Phase II clinical trial of SHR-A1811 for injection in patients with HER2-expressing recurrent or metastatic cervical cancer who have failed prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study, sign the informed consent, have good compliance, and can cooperate with follow-up.
2. Female, aged 18-75 years old (including 18 and 75 years old, calculated on the day of signing the informed consent).
3. Cervical cancer confirmed by tissue or cytological pathology.
4. Expected survival ≥ 12 weeks.
5. Normal function of important organs.
6. Female subjects of fertility must have a negative serum HCG test within 7 days before the first dose of Investigational Medicinal Product (IMP), and must not be breastfeeding, and must agree to comply with contraceptive requirements from the signing of the informed consent until the last dose of the trial drug for 7 months.

Exclusion Criteria:

1. Subjects with known untreated or active central nervous system (CNS) tumor metastases.
2. Subjects with other malignant tumors in the past or at the same time.
3. Subjects with clinically symptomatic, poorly controlled, or moderate or greater pleural effusion, pericardial effusion or peritoneal effusion.
4. Subjects with a history of interstitial pneumonia/interstitial lung disease or non-infectious pneumonia requiring steroid treatment.
5. Subjects with autoimmune, connective tissue or inflammatory diseases involving the lungs.
6. Subjects with known lung damage caused by concurrent lung diseases.
7. Subjects with active pulmonary tuberculosis.
8. Subjects with poorly controlled or severe cardiovascular diseases.
9. Subjects with arterial/venous thrombotic events within 1 month before enrollment.
10. Subjects who had a serious infection within 1 month before enrollment.
11. History of immunodeficiency, including positive HIV test.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by Independent Review Committee (IRC) | Up to 2 years.

SECONDARY OUTCOMES:
Overall survival (OS) assessed by Independent Review Committee (IRC) | Up to 2 years.
Overall survival (OS) assessed by investigators | Up to 2 years.
Progression free survival (PFS) assessed by Independent Review Committee (IRC) | Up to 2 years.
Progression free survival (PFS) assessed by investigators | Up to 2 years.
Duration of response (DoR) assessed by Independent Review Committee (IRC) | Up to 2 years.
Duration of response (DoR) assessed by investigators | Up to 2 years.
Disease control rate (DCR) assessed by Independent Review Committee (IRC) | Up to 2 years.
Disease control rate (DCR) assessed by investigators | Up to 2 years.
Objective response rate (ORR) assessed by investigators | Up to 2 years.
Adverse events (AEs) | Up to 2 years.
Serious adverse events (SAEs) | Up to 2 years.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Shandong University Qilu Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided